CLINICAL TRIAL: NCT06188273
Title: Impact of Skeletal Muscle Quality and Loss on the Outcome of Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Shulan (Hangzhou) Hospital (Other); The Affiliated Hospital of Qingdao University (Other); West China Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2023-ZJU-OBS3
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplantation; Muscle Loss; Muscle Quality
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Myosteatotic Group: The group of patients was diagnosed with myosteatosis through CT imaging assessment before transplantation.
- Non-myosteatotic Group: The group of patients was diagnosed without myosteatosis through CT imaging assessment before transplantation.
- The Group with Severe Muscle Loss: The group of patients, through the comparison of CT images before and after transplantation, was diagnosed with significant muscle loss.
- The Group without Severe Muscle Loss: The group of patients, through the comparison of CT images before and after transplantation, was diagnosed without significant muscle loss.

SUMMARY:
CT imaging-based skeletal muscle assessment has been found to predict the outcomes of many diseases. Previous evidence revealed that pre-transplant muscle quality and post-transplant muscle loss were associated with transplant outcomes. However, there is no prospective study supporting the aforementioned conclusions. This study aims to prospectively include liver transplant patients from multiple transplant centers, collecting their pre-transplant CT images as well as post-transplant CT images at specific time points. The objective is to further explore and clarify the correlation between skeletal muscle assessment and the prognosis of liver transplant patients. The goal is to provide guidance for peri-transplant health monitoring and disease intervention for liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing deceased donor liver transplantation (DDLT) for the first time

Exclusion Criteria:

* Pediatric transplants
* Presence of portal vein tumor thrombus according to imageing before transplantation
* Presence of macrovascular invasion according to imageing before transplantation
* Re-transplants
* Multi-organ transplants
* Patients who died within 30 days after transplantation
* Patients diagnosed with skeletal muscle diseases (e.g. muscle atrophy)
* Patients with serious medical conditions such as heart failure, persistent infection, and renal insufficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant patients from multiple transplant centers in China
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative mortality | 2024.1.1-2027.1.1
Postoperative recurrence of liver cancer | 2024.1.1-2027.1.1
  Specifically for the included patients who undergo liver transplantation for liver cancer